CLINICAL TRIAL: NCT05335863
Title: Clinical Trial to Evaluate Hypercaloric/High-protein Nutritional Supplement Glycemic Index Enriched With Calcium, Vitamin D and Docosahexaenoic Acid (DHA) in Healthy Adults
Brief Title: Glycemic Index Evaluation of a Hypercaloric/High-protein Nutritional Supplement in Healthy Adults
Acronym: TERATROFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Fundacio Eurecat (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HULP 5921
Record Dates: First submitted 2021-07-18; First posted 2022-04-20 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: diabetes; oral nutritional supplement; glycemic index; healthy population
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dietary Supplements; Glucose

STUDY DESIGN:
Intervention Model Description: Crossed, controlled and randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Ingestion of FontActiv® DiaBest high protein/hypercaloric
  Interventions: Dietary Supplement: Oral Nutritional Supplement
- Control (Placebo Comparator): Ingestion of glucose standard solution
  Interventions: Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplement — Participants must consume 416 mL of ONS FontActiv® DiaBest HP / HC vanilla flavor. A maximum time of 10 min will be given to consume the entire product.
  Other Names: Experimental
  Arms: Experimental
Dietary Supplement: Glucose — Participants must consume a 50 g glucose solution in 10 min to obtain the ares under the curve (AUC) data from glucose consumption
  Arms: Control

SUMMARY:
Diabetes mellitus (DM) is a chronic disease with a higher prevalence in the world population, especially in the elderly population.The main consequence of the alteration of DM is the increase in blood glucose levels. When the concentration reaches levels above 180-200 mg / dl after ingestion, the following symptoms appear: polyphagia, polydipsia, polyuria and weight loss. Diet, on some occasions, is the only therapy necessary. The commercialized formulas considered as "standard", have a high content of carbohydrates with a high glycemic index (approximately 50%) and low in lipids (30-35%) and do not usually contain fiber. This type of liquid formulations seem to increase the insulin and glycemic response in healthy people, and to a greater extent in patients with DM, compared to what would cause a similar intake of nutrients in a mixed diet.

All diabetic formulas provide carbohydrates with low glycemic index. They are made from starches, with a variable contribution of fructose, which in all cases should be less than 20% of the total caloric intake, due to its lower glycemic index, its greater sweetening power and its entry into the cell is insulin-independent. However, it is necessary to determine the glycemic index of the new specific formulas for this population through clinical trials.Based on these initial facts, researchers consider it appropriate to carry out a pilot study to evaluate the glycemic index of a Oral Nutritional Supplement (ONS) especially indicated for diabetic people in a group of healthy people.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic disease with a higher prevalence in the world population, especially in the elderly population. It is considered one of the main health problems worldwide. Taking into account the aging of the population, the increase in obesity and the sedentary lifestyle, the World Health Organization (WHO) predicts that disease incidence in developed countries will increase. In Spain, DM affects 6% of the population; being more frequent type 2 DM in the elderly population. Nearby 20% of the Spanish population> 60 years of age suffers from it. In type 2 DM there is resistance to insulin, in addition to a deficit in its production. Concerning hyperglycemia, both phenomena must be present.

The main consequence of the alteration of DM is the increase in blood glucose levels. When the concentration reaches levels above 180-200 mg / dL after ingestion, the following symptoms appear: polyphagia, polydipsia, polyuria and weight loss. These short-term symptoms are the most common. Diabetes prevention is based on an integrated holistic approach based on healthy eating, daily physical exercise and adequate health education. To achieve a proper balance between these three pillars, patient collaboration is required.

Most of cases just need diet as the only therapy needed. The importance of weight loss is highlighted, since approximately 80% of patients with DM 2 have a BMI> 25 kg / m2. The main objective of the diet is to achieve normal blood glucose levels both in the fasting state and in the postprandial phase. Blood pressure and lipid control are also important. However, elderly diabetic patients are more likely to suffer from malnutrition associated with the disease, with a higher prevalence than in the general population. The prevalence of the diabetic patient referring to the hospital setting ranges between 5-11%. However, extracted data from hospital discharges rise up to 20%, if medical records are considered.

The main indications for enteral nutrition (EN) application, according to data from 2001, were neurological alterations (43.3%) and neoplasms (39%), which are frequent pathologies in elderly patients. Regarding hospitalized patients, between 5-10% receive some type of nutritional support. When prevalence rate of diabetic patients is applied to this population group, 1-2% of hospitalized diabetic patients are prescribed with some type of nutritional supplement. Malnutrition in diabetic patients worsens if the supplements are not correctly tolerated, leading to a worse diagnosis due to the difficulty in healing and the greater propensity for infections, leading to longer hospital stays.

The commercialized formulas considered as "standard", have a high content of carbohydrates with a high glycemic index (approximately 50%) and low lipids (30-35%) and do not usually contain fiber. This type of liquid formulations seems to increase the insulin and glycemic response in healthy people, and to a greater extent in patients with DM, compared to what would cause a similar intake of nutrients in a mixed diet. It seems that when ingesting a formula with a low carbohydrate content and high content of monounsaturated fatty acids, the postprandial glycemic response depends fundamentally on the total carbohydrate content, downplaying the source (starch or fructose) or even the addition or type of fiber. Therefore, it seems that as the carbohydrate content increases, the lipid content could contribute to the attenuation of the glycemic response. However, more comparisons are needed between specific diabetes diets (high, moderate, and low fat) with each other and with other standard diets (with and without fiber).

All diabetic formulas provide carbohydrates with low glycemic index. They are made from starches, with a variable contribution of fructose. Fructose should be less than 20% of the total caloric intake in all cases, due to its lower glycemic index, its greater sweetening power and its entry into the cell as insulin-independent. However, it is necessary to determine the glycemic index of the new specific formulas for this population through clinical trials.

Based on these initial facts, researchers consider to carry out a pilot study to evaluate the glycemic index of a Oral Nutritional Supplement (ONS) especially indicated for diabetic patients in a group of healthy people.

ELIGIBILITY:
INCLUSION CRITERIA

* Men and women between 18 and 65 years
* Patients without chronic uncontrolled diseases
* Patients willing to consume the Oral Nutritional Supplement (ONS) to carry out the study
* Patients with adequate cultural level and understanding of the clinical study
* Patients who agree to voluntarily participate in the study and who give their informed consent in writing

EXCLUSION CRITERIA

* Subjects with any serious chronic pathology.
* Subjects with metabolic or intestinal pathologies that interfere with the homeostatic mechanisms of glucose
* Subjects with neurological pathologies or eating disorders that interfere with acute tests.
* Subjects with allergies or intolerances to any of the ingredients in the formula
* Subjects with socio-family problems that prevent them from participating in the study
* Subjects with intense physical activity
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Areas under the glucose metabolism curve for the determination of the glycemic index | 0-120 minutes
  Statistical calculation of the area under the curve at different times of blood collection (baseline, 0, 30, 60, 90 and 120 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Bricia López-Plaza, MsC, PhD, Principal Investigator — Instituto de Investigación Hospital Universitario La Paz
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No